CLINICAL TRIAL: NCT06289959
Title: A Prospective, Single-Center, Randomized, Controlled Study Guiding the Treatment of Diffuse Large B-Cell Lymphoma Patients Based on Plasma cfDNA Testing
Brief Title: Plasma cfDNA Testing Guiding the Treatment Decisions of DLBCL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JD-LC2023006-I01
Record Dates: First submitted 2024-01-25; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: cfDNA; therapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group1（Plasma cfDNA-negative patients） (Active Comparator): Continue to receive monotherapy with rituximab （375mg/m2 q3w）for 2 cycles
  Interventions: Diagnostic Test: cfDNA
- Group2（plasma cfDNA-positive patients） (Experimental): Continue monotherapy with rituximab （375mg/m2 q3w）for 2 cycles
  Interventions: Diagnostic Test: cfDNA
- Group3（plasma cfDNA-positive patients） (Experimental): Receive the original regimen for 2 cycles（R-CHOP like）
  Interventions: Diagnostic Test: cfDNA

INTERVENTIONS:
Diagnostic Test: cfDNA — After achieving complete metabolic remission (Lugano response assessment criteria) following 6 cycles of R-CHOP-like chemotherapy, patients undergo plasma cfDNA testing upon enrollment，and the follow-up treatment plans are based on cfDNA results.

SUMMARY:
A prospective, single center, randomized, clinical controlled study to evaluate the efficacy and prognosis differences between precision treatment based on plasma cfDNA testing results and the current conventional diagnostic and treatment practices for DLBCL patients.

DETAILED DESCRIPTION:
This study is initiated by researchers and is a prospective, single-center, randomized, clinical controlled study. The study subjects are newly diagnosed DLBCL patients with plasma cfDNA positivity (defined as positive for point mutations, CNV, IgH-related fusion, or IG clonal rearrangement). After achieving complete metabolic remission (Lugano response assessment criteria) following 6 cycles of R-CHOP-like chemotherapy, patients undergo plasma cfDNA testing upon enrollment. Plasma cfDNA-negative patients (Group 1) continue to receive monotherapy with rituximab for 2 cycles, while plasma cfDNA-positive patients are randomly assigned to Group 2 and Group 3. Group 2 patients continue monotherapy with rituximab for 2 cycles, and Group 3 patients receive the original regimen for 2 cycles. Plasma cfDNA testing is performed again for all three groups after completion of the entire treatment. Patient progression-free survival (PFS) is observed for 2 years. After treatment completion, follow-up visits are scheduled every 3 months for a total of 24 months.

Research Objective: Evaluate the efficacy and prognosis differences between precision treatment based on plasma cfDNA testing results and the current conventional diagnostic and treatment practices for DLBCL patients.

Expected Results: Determining subsequent treatment based on plasma cfDNA MRD results at the end of DLBCL patient treatment is expected to aid in identifying high-risk patients for early relapse and improving their prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, gender not specified.
* Newly diagnosed patients with diffuse large B-cell lymphoma (DLBCL) confirmed by histopathological examination. Patients should test positive for plasma cfDNA before treatment (defined as positive for point mutations, CNV, IgH-related fusion, or IG clonal rearrangement) and achieve complete metabolic remission after 6 cycles of R-CHOP chemotherapy (evaluated by Lugano response assessment criteria).
* Patients for whom the researcher predicts a life expectancy of >6 months.
* Signed informed consent form.

Exclusion Criteria:

* Patients who have undergone autologous stem cell transplantation.
* Patients with a history of other malignant tumors, except for basal cell carcinoma of the skin or in situ cervical cancer.
* Patients with uncontrolled cardiovascular diseases, coagulation disorders, connective tissue diseases, severe infectious diseases, and other such conditions;
* Primary central nervous system lymphoma.
* Patients with mental illness or others known or suspected to be unable to fully comply with the study protocol.
* Pregnant or lactating women.
* HbsAg-positive patients who need to undergo HBV-DNA testing and can only be included if they seroconvert. Additionally, if the HbsAg test is negative but the HBcAb test is positive (regardless of HbsAb status), HBV-DNA testing is also required. If the result is positive, inclusion is possible only after seroconversion.
* HIV-infected individuals.
* Other concurrent and uncontrolled diseases that researchers believe may affect the medical condition of patients participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-25 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival（PFS） | From date of randomization until the date of first documented progression or date of death from any cause,whichever came first，assessed up to 24 months.
  Evaluate the PFS among three groups with different treatment practices for diffuse large B-cell lymphoma (DLBCL) patients.

SECONDARY OUTCOMES:
Sensitivity, and specificity of plasma cfDNA in DLBCL patients | From date of randomization until the date of first documented progression or date of death from any cause,whichever came first，assessed up to 24 months.
  Evaluate the sensitivity, and specificity of plasma cfDNA testing at the end of treatment in DLBCL
Overall survivals(OS) | From date of randomization until the date of first documented progression or date of death from any cause,whichever came first，assessed up to 24 months.
  overall survival in DLBCL patients.

CONTACTS AND LOCATIONS:
Overall Officials: Bingzong Li, Professor, Study Chair — Second Affiliated Hospital of Soochow University
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No